CLINICAL TRIAL: NCT04372641
Title: A Phase I Trial of the P97 Inhibitor CB-5339 in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: Testing the Safety of CB-5339 in Patients With Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Clinical development of the agent has been discontinued
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08664; NCI-2019-08664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10349 (Other: National Cancer Institute LAO); 10349 (Other: CTEP); NCT04449562 (obsolete NCT alias)
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; Indolent Non-Hodgkin Lymphoma; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (p97 inhibitor CB-5339 tosylate) (Experimental): Patients receive p97 inhibitor CB-5339 tosylate PO QD 4 days on and 3 days off. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: p97 Inhibitor CB-5339 Tosylate

INTERVENTIONS:
Drug: p97 Inhibitor CB-5339 Tosylate — Given PO
  Other Names: CB 5339 Tosylate; CB-5339 Tosylate; CB5339 Tosylate

SUMMARY:
This phase I trial studies the side effects and best dose of CB-5339 in treating patients with solid tumors that has spread to other places in the body (advanced) or lymphomas. CB-5339 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety, tolerability, and recommended phase 2 dose (RP2D) of p97 inhibitor CB-5339 tosylate (CB-5339) administered orally on a schedule of once daily, 4 days on and 3 days off, in patients with advanced solid tumors and lymphomas.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic profiles of CB-5339. II. To assess the preliminary antitumor activity of CB-5339 in patients with advanced solid tumors and lymphomas.

III. To determine the effects of CB-5339 on the ubiquitin proteasome system and on markers of cell death in pre- and post-treatment tumor biopsies and peripheral blood mononuclear cell (PBMC)s.

EXPLORATORY OBJECTIVE:

I. To evaluate potential associations between CB-5339 activity and genomic alterations assessed in circulating tumor deoxyribonucleic acid (DNA) (ctDNA).

OUTLINE: This is a dose-escalation study.

Patients receive p97 inhibitor CB-5339 tosylate orally (PO) once daily (QD) 4 days on and 3 days off. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented metastatic or locally advanced (not amenable to surgery) solid tumors whose disease has progressed on standard therapy or for which there is no available standard therapy or therapy known to prolong survival; or aggressive lymphoma who have refused or have no remaining curative options (e.g., stem cell transplant). Patients with indolent lymphomas must have undergone 3 or more prior regimens of therapy
* Any prior therapy must have been completed >= 4 weeks (6 weeks for nitrosoureas and mitomycin C) or, if known, >= 5 half-lives of the prior agent (whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment), and the participant must have recovered to eligibility levels from prior toxicity. Prior definitive radiation should have been completed >= 4 weeks or palliative radiation should have been completed >= 2 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels (patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the principal investigator [PI]'s discretion). Patients must be >= 2 weeks since any investigational agent administered as part of a phase 0 study (where a sub-therapeutic dose of drug is administered) at the PI's discretion and should have recovered to grade 1 or baseline from any toxicities
* Patients who have had prior monoclonal antibody therapy must have completed that therapy >= 6 weeks (or 3 half-lives of the antibody, whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%) and life expectancy > 3 months
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL (solid tumor patients)
* Platelets >= 75,000/mcL (lymphoma patients)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR 60 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 x institutional normal
* The effects of CB-5339 on the developing human fetus are unknown. For this reason and because p97 inhibitors agents may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 4 months afterwards. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CB-5339 administration
* Ability to understand and the willingness to sign a written informed consent document
* Subjects on the expansion cohort must also be willing to undergo two core biopsy procedures if there is a lesion amenable to biopsy
* Left ventricular ejection fraction >= the lower limit of normal by echocardiogram (ECHO) at entry
* Mean QT interval corrected for heart rate (QTc) < 470 ms using Fridericia's correction

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with clinically significant illnesses which would compromise participation in the study, including but not limited to active or uncontrolled infection, immune deficiencies, hepatitis B, hepatitis C, active tuberculosis, uncontrolled asthma, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, myocardial infarction within the past 6 months, cerebral vascular accident/stroke within the past 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.

  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for >= 4 weeks after treatment of the brain metastases. Patients on anti-seizure medications may be enrolled at the discretion of the principal investigator providing that these patients are taking non-enzyme- inducing anti-seizure medications or can be converted to these
* Pregnant women are excluded from this study because CB-5339 may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with this agent, breastfeeding should be discontinued if the mother is treated with CB-5339
* Current or previous history of sight-threatening retinal disease, including (but not limited to) proliferative diabetic retinopathy, severe retinal vascular disease, and advanced age-related macular degeneration
* Patients with a history of QT-prolongation or of Torsades de pointes (TdP), or of taking QT-prolonging drugs, are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-18 (Estimated); Primary Completion 2021-07-12 (Estimated); Study Completion 2021-07-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase I) | 30 days
Recommended phase II dose (Phase I) | 30 days

SECONDARY OUTCOMES:
Pharmacodynamic analysis (expansion phase) | Up to 2 years
Response assessment | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Naoko Takebe, Principal Investigator — National Cancer Institute LAO
Locations (2):
- United States (2):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT04372641/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04372641/ICF_001.pdf